CLINICAL TRIAL: NCT01564160
Title: Assessment of the Acute and Chronic Bioavailability of Marine Lipid Fraction PCSO-524 Relative to a Comparator Product.
Brief Title: Assessment of PCSO-524 Relative to a Comparator Product
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Nutrasource Pharmaceutical and Nutraceutical Services, Inc. (Network)
Collaborators: Pharmalink International Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 11.0202; 176412 (Other: Health Canada); 12-02-003 (Other: Canadian SHIELD Ethics Review Board)
Record Dates: First submitted 2012-03-22; First posted 2012-03-27 (Estimated); Last update posted 2012-12-03 (Estimated); Status verified 2012-11

CONDITIONS: Healthy
Keywords: Fish Oil; EPA; DHA; Omega-Score; Omega-3 Fatty Acids; Green-Lipped Mussel; Omega-score < 5.2%
MeSH Terms: interventions — Fish Oils; PCSO-524

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1: PCSO-524 (Experimental): PCSO-524
  Interventions: Dietary Supplement: PCSO-524
- Arm 2: Fish Oil (Active Comparator): Fish Oil
  Interventions: Dietary Supplement: Fish Oil

INTERVENTIONS:
Dietary Supplement: Fish Oil — Source of omega-3 fatty acids.
  Arms: Arm 2: Fish Oil
Dietary Supplement: PCSO-524 — Extract of Greenshell Mussel
  Arms: Arm 1: PCSO-524

SUMMARY:
A marine lipid oil extract isolated from the New Zealand Greenshell® Mussel, Perna canaliculus (P. canaliculus), contains a unique synergistic blend of marine fatty acids.

The objective of the this study is to evaluate the acute (5-hour) and chronic (21-day) bioavailability of a fixed dose of PCSO-524 compared to a fish oil product in a population of healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* The individual is fluent in English and understands the study requirements
* The participant is willing and able to comply with all requirements defined within this protocol.
* The individual is willing to provide written informed consent
* The individual is male or female
* The individual is between 18 and 65 years of age
* The individual's blood EPA+DPA+DHA ≤ 5.2% at screening

Exclusion Criteria:

* The individual is unable to or refuses to provide written informed consent
* The individual has taken omega-3 supplements within 3 months of screening.
* Supplements containing any of the following sources of omega-3s will exclude the individual from the study: fish oil, flax oil, krill oil, green-lipped mussel, chia, perilla, algea
* The individual's blood EPA+DPA+DHA ≥ 5.2% at screening
* The individual is female and pregnant or breastfeeding, or plans to be during the trial period
* The individual has known allergies product ingredients (fish/seafood)
* The individual has any significant medical illness or condition
* The individual has reported a history of drug dependence or substance abuse (excluding nicotine)
* The individual is taking lipid-altering medications (statins, niacin, carnitine, fibrates etc.)
* The individual is unable to abstain from caffeine, alcohol or physical activity for 24 hours before each treatment visit
* The individual will be excluded if he or she has any additional conditions that, in the Investigator's opinion, would preclude the participant from completing the study or would not be in the best interest of the subject. This would include any significant illness or unstable medical condition that could lead to difficulty complying with the protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2012-04; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Serum Phospholipid | Day 0 and Day 21

SECONDARY OUTCOMES:
Total Serum Lipid | Day 21 @ 0 hours, 2 hours, 3 hours, 4 hours and 5 hours post-dose
Serum Free Fatty Acid | Day 21 @ 0 hours, 2 hours, 3 hours, 4 hours and 5 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Maggie D Laidlaw, Ph.D, Principal Investigator — Nutrasource Diagnostics
Locations (1):
- Nutrasource Diagnostics Inc, Guelph, Ontario, Canada